CLINICAL TRIAL: NCT06395688
Title: A Double Blind, Placebo-controlled Trial in Healthy Volunteers to Investigate the Effect of Multiple Oral Doses of AEF0117 Versus Placebo on the Pharmacokinetics of THC and Its Metabolites 11 OH THC and THC COOH When Smoking Cannabis.
Brief Title: Drug-Drug Interaction Between THC and AEF0117
Acronym: DDI
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aelis Farma (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEF0117-107; U01DA053832 (NIH)
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Cannabis Abuse
Keywords: Cannabis use disorder
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AEF0117 (Experimental): Participant will be administered once daily 2 placebo capsules for 1 day and 2 AEF0117 capsules for 7days
  Interventions: Drug: 3ß-(4-methoxybenzyloxy)pregn-5-en-20-one; Drug: Placebo
- Placebo (Placebo Comparator): Participant will be administered once daily 2 placebo capsules for 8 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 3ß-(4-methoxybenzyloxy)pregn-5-en-20-one — AEF0117 soft capsules of 1mg
  Other Names: AEF0117
  Arms: AEF0117
Drug: Placebo — Placebo soft capsules (identical to active compound)

SUMMARY:
This trial is a single center, double blind, placebo-controlled trial in healthy male and female recreational cannabis users with placebo and AEF0117 dosed in a fixed sequence.

The goal of this clinical trial is to investigate if AEF0117 has any effect on the pharmacokinetics of THC and its metabolites when smoking cannabis.

DETAILED DESCRIPTION:
The goal of this clinical trial is to investigate if AEF0117 has any effect on the pharmacokinetics of THC and its metabolites when smoking cannabis.

Participants will be male or female in good health aged from 21y to 55y old and who are recreational cannabis users.

The participant will receive either AEF0117 (2 mg) or placebo. The sponsor team, the research staff and the participant won't know which study medication has been given.

The main objectives of the trial are:

* To compare the effect of AEF0117 multiple doses on the maximal plasma concentration and other pharmacokinetic parameters of the THC and its metabolites.
* To investigate safety and tolerability of multiple doses of AEF0117 and when co-administered with a dose of smoked cannabis.

The participant will come for 2 inpatient phases (including one overnight stay). Those 2 inpatient phases are separated by 5 days at home.

After a screening period assessing the good health and the eligibility of the participant, on day 1 they will receive 2 capsules of the study medication and will smoke one cannabis cigarette. During the day, blood samples will be collected at defined timepoints before the study medication, after the study medication and before smoking and after smoking.

On day 2, Blood samples will be collected before and after the study medication intake.

At the end of the assessements, the participant will be discharged. They could be requested to stay at the research facility if they experience any adverse effects From Day 3 to Day 7, the participant will be contacted by phone or by videoconference to confirm the study medication intake and if they experience any adverse events.

On day 8, the participant will come back to the research facility for a 2 days visit including an overnight stay. Assessments and procedures will similar to those performed on Day 1 and Day 2.

On Day 14, the participant will come back to the research facility a last time for a final blood collection.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females of any race, 21 to 55 years old, both inclusive.
2. Subjects must use highly effective contraception.

   * Participants who engage in heterosexual sex must use highly effective contraception during the entire trial period. Male participants should refrain from donating sperm or planning a pregnancy throughout the trial. Female participants who are heterosexually active are eligible if: they use highly effective contraception or are post-menopausal and with a negative pregnancy test. Use of hormonal contraception must have been stable for 3 months prior to screening and expected to be unchanged during the trial.
3. Body mass index (BMI) between 20.0 and ≤35.0 kg/m2 at screening.
4. Be informed of the nature of the trial and provide written informed consent.
5. Be legally competent and able to communicate effectively (in English) with trial personnel.
6. Cannabis smoker (use ≥1 day the last 2 months and ≤2 days/week) who agrees to abstain from cannabis (except for what is provided by investigators) for 3 days prior to and including Day 1 and Day 8 of the study, and while in the clinic.

Exclusion Criteria:

1. Severe learning disability, brain damage, or pervasive developmental disorder.
2. Any disease or condition that according to the investigator's medical judgment might compromise the cardiovascular, hematologic, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) systems.
3. Any clinical laboratory values assessed as clinically significant by the investigator.
4. a) A history of alcohol- or substance use disorders within the past 2 years, recent or current regular use of any illicit drugs except cannabis. In case of a positive drug screen (except for cannabis) at screening, a negative test is required at re-screening.

   b) The alcohol breath test and urine drug screen at predose Day 1 must be negative (including for cannabis, a level of THC-COOH <100 ng/mL is allowed).
5. A history of or current serious mental illness including active or recent suicidal ideation, severe psychological distress (e.g., active suicidal plans, psychosis, debilitating panic disorder), and/or an abnormal Columbia-Suicide Severity Rating Scale (C-SSRS) result (i.e., a C-SSRS score of ≥3).
6. History of COVID-19 within 4 weeks prior to Day 1, or positive COVID 19 test if required according to standard procedures at the site.
7. A history of difficulty donating blood or inadequate venous access.
8. Blood pressure outside normal range (140/80 mmHg systolic/diastolic) and considered potentially clinically significant by the investigator.
9. A corrected QT interval (Fridericia's correction, QTcF) >450 msec for males and >470 msec for females.
10. Clinically significant anemia or low hemoglobin (levels <9 g/dL) at screening, donation of >250 mL of blood or plasma or received any blood and plasma for medical/surgical reasons within the 30 days prior to receiving trial drug, or intention to donate blood or plasma within 1 month after receiving trial drug.
11. Allergies to the trial drug and known allergies to corn or corn derivatives.
12. Use of any prescription or over-the-counter drug therapy, including psychoactive and/or psychotropic medication, herbal or homeopathic supplements unapproved by the sponsor within 2 weeks prior to receiving the trial drug (for drugs with an elimination half-life greater than 10 days, this will be extended to 60 days).
13. Use of bodybuilding supplements, any food supplement or topical product containing pregnenolone, or any other steroid, including phytosteroids.
14. Use of a diet or supplements (e.g., St. John's Wort), or food and fruit juices (e.g., grapefruit juice, Sevilla oranges) known to induce or inhibit hepatic drug metabolism within 2 weeks prior to receiving the trial drug and until the follow-up visit, unless approved by the sponsor's medical monitor.
15. Tobacco smokers who smoke more than 5 cigarettes per day or use an equivalent daily amount of other tobacco products and are not willing to abstain from tobacco smoking during the inpatient visits.
16. Legal status that would interfere with participation.
17. Unable to follow the restrictions outlined in the protocol.
18. Use of an investigational drug or product, or participation in a drug trial within the last 90 days prior to receiving the trial drug.
19. Participation in a previous trial with AEF0117 within the last 3 months prior to screening.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Cmax for co-administration of THC and AEF0117 | Day1, Day8
  Comparison of the maximal plasma concentration (Cmax) of THC after co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo.

SECONDARY OUTCOMES:
AUC for co-administration of THC and AEF0117 | Day1, Day8
  Comparison of the area under the curve (AUC) of THC after co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo.
Tmax for co-administration of THC and AEF0117 | Day1, Day8
  Comparison of time of peak concentration of THC after co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo
Tlag for co-administration of THC and AEF0117 | Day1, Day8
  Comparison of Tlag of THC after co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo
Clast for co-administration of THC and AEF0117 | Day1, Day8
  Comparison of Clast of THC after co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo
t1/2 for co-administration of THC and AEF0117 | Day1, Day8
  Comparison of plasma half-life (t1/2) of THC after co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo
Cmax for 11-OH-THC and THC-COOH | Day1, Day8
  Comparison of peak concentration (Cmax) of 11-OH-THC and THC-COOH after co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo
AUC for 11-OH-THC and THC-COOH | Day1, Day8
  Comparison of the area under the curve (AUC) of 11-OH-THC and THC-COOH after co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo
Tmax for 11-OH-THC and THC-COOH | Day1, Day8
  Comparison of the time of peak concentration (Tmax) of 11-OH-THC and THC-COOH after co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo
Tlag for 11-OH-THC and THC-COOH | Day1, Day8
  Comparison of Tlag of 11-OH-THC and THC-COOH after co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo
Incidence of TEAEs or TESAEs | From Day1 to Day14
  Assessed by AE and SAE reporting
Incidence of TEAEs and TESAEs assessed by vital signs | Day1, Day2, Day8, Day9, Day14
  By evaluating changes from the baseline in vital signs
Effect on heart rate | Day1, Day8
  Measurement of Heart rate over predefined time intervals from prior to IMP dosing until 11 hours after dosing during co-administration of cannabis cigarette and AEF0117 versus co-administration of cannabis cigarette and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, PhD, Principal Investigator — New York Institute Psychiatric Institute

IPD SHARING:
Plan to Share IPD: No